CLINICAL TRIAL: NCT06699953
Title: Characterizing the EEG Signature of Fentanyl and Its Association With Drug Liking
Status: Enrolling by invitation | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Patrick Purdon, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Other Study IDs: IRB-77223; R01DA056593 (NIH)
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Brain Activity Related to Opioid Administration; Brain Activity Related to Drug Liking
Keywords: opioid crisis; neuroscience; EEG; drug liking; fentanyl; anesthesia; general anesthesia; opioids; analgesia
MeSH Terms: conditions — Agnosia | interventions — Observation; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study in patients receiving fentanyl for surgery — This observational study enrolls patients receiving fentanyl, a drug routinely administered during surgery under general anesthesia. The primary difference in the investigators' research protocol is the inclusion of a 5-minute interval between fentanyl administration and the induction of general anesthesia. Fentanyl will be given in two boluses of 2 mcg/kg (ideal body weight), spaced 2 minutes apart, totaling 4 mcg/kg. If the participant remains conscious, an additional 2 mcg/kg bolus will be administered after 2 minutes. Additionally, participants will complete a drug-liking questionnaire before the first bolus and every 30 seconds until anesthesia induction, rating how much they "liked" the drug on a 0-100 scale.

SUMMARY:
The goal of this study is to characterize an electroencephalogram (EEG) biomarker for fentanyl and understand where this signal is coming from in the brain. The investigators also aim to understand how this EEG biomarker is connected to patient perception to drug liking.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or above (male and female)
2. American Society of Anesthesiologists (ASA) physical status classification of I, II or III
3. Candidates scheduled for general surgical procedures under general anesthesia and receive fentanyl for surgery

Exclusion Criteria:

1. Craniofacial abnormalities
2. Known or suspected difficult intubation or mask ventilation
3. Known or suspected need for rapid sequence induction and intubation
4. Body mass index above 45 kg/m2
5. Allergies to fentanyl
6. History of obstructive sleep apnea requiring CPAP
7. History of obstructive or restrictive lung disease
8. Opiate use within 24 hours
9. History of opiate abuse within the last 3 years
10. Known or suspected severe chronic pain condition that require use of opiates or limit daily activities
11. MRI contraindications, such as presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, or body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for general surgical procedures under general anesthesia
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Source Localization of Fentanyl EEG Signature | 15 minutes prior to surgery
  The investigators will perform high density electroencephalogram to estimate the power and source localization of canonical (delta, theta, alpha, gamma and beta) bands power to determine the likely generators for the fentanyl EEG signature.

SECONDARY OUTCOMES:
Relationship Between Fentanyl EEG Signature and Fentanyl Effect Site Concentration | 15 minutes prior to surgery
  The investigators will use a linear mixed-effects model to characterize the relationship between the fentanyl EEG signature and fentanyl predicted effect site concentrations derived from pharmacokinetic models.
Relationship Between Visual Analog Scale Liking Rating and Fentanyl EEG Signature | 15 minutes before the surgery
  The investigators will use a linear mixed-effects model to characterize the relationship between the VAS (0 - 100) liking rating and the fentanyl EEG signature.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balanza GA, Bharadwaj KM, Mullen AC, Beck AM, Work EC, McGovern FJ, Houle TT, Eric TP, Purdon PL. An electroencephalogram biomarker of fentanyl drug effects. PNAS Nexus. 2022 Aug 30;1(4):pgac158. doi: 10.1093/pnasnexus/pgac158. eCollection 2022 Sep. PMID 36329725